CLINICAL TRIAL: NCT00306930
Title: Multi-center, Prospective, Clinical Evaluation of Pinnacle Acetabular Implants in Total Hip Arthroplasty
Brief Title: Clinical Study Evaluating an Acetabular Cup System After Total Hip Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIN
Record Dates: First submitted 2006-03-23; First posted 2006-03-27 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Arthritis; Avascular Necrosis; Acute Fracture
Keywords: Total Hip Replacement; post-traumatic arthritis
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Arthritis; Osteonecrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Other): Acetabular cup replacement with total hip arthroplasty
  Interventions: Device: Acetabular cup

INTERVENTIONS:
Device: Acetabular cup — Acetabular cup replacement
  Other Names: Pinnacle™ Cup

SUMMARY:
This study is a clinical evaluation of survivorship of an acetabular cup system after total hip replacement using patient examinations and questionnaires.

DETAILED DESCRIPTION:
The primary objective of this investigation is to evaluate survivorship at five years of the Pinnacle™ acetabular cup system in primary total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Primary hip replacement
* Sufficient bone stock to support implant
* Signed Informed Patient Consent form

Exclusion Criteria:

* Prior renal transplant
* History of active joint sepsis
* Recent high dose of corticosteroids
* Primary or secondary carcinoma in the last 5 years
* Neurological disease
* Psychosocial disease that would limit rehabilitation
* Use of structural bone graft
* Simultaneous participation in another hip study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1593 (Actual)
Dates: Start 2000-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Survivorship | 5 years

SECONDARY OUTCOMES:
Harris Hip Score | Pre-operative, 6 month and 1, 2, 3, 4, and 5 years.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Pre-operative, 6 month and 1, 2, 3, 4 and 5 years.
Short Form-36 (SF-36) | Pre-operative, 6 month and 1, 2, 3, 4 and 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Dave Whalen, BS, DC, Study Director — DePuy Orthopaedics
Locations (1):
- DePuy Orthopaedics, Warsaw, Indiana, United States